CLINICAL TRIAL: NCT03346382
Title: Treatment of Epilepsy in Children and Adults in the Emergency Medical Services of the City of Zurich, Switzerland - Midazolam Versus Diazepam - A Retrospective Analysis
Brief Title: Emergency Medical Services and Epilepsy in Switzerland
Status: Completed | Type: Observational
Sponsor: Theusinger Oliver M. (Other)
Responsible Party: Sponsor-Investigator, Theusinger Oliver M., Principal Investigator, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Other Study IDs: OMT 01012015 SRZ
Record Dates: First submitted 2017-11-02; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
Keywords: Epilepsy; Emergency medical services
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective data analysis, all emergency medical services of the city of Zurich interventions due to epileptic convulsions during June 2013 and December 2014 have been analyzed regarding the type of drug used, its application mode and the application mode based success. Furthermore, children versus adults were compared. Continuous variables were summarized as mean ± standard deviation (SD) and also presented as median [minimum; maximum]. Groups were compared using the independent samples t-test. P-values < 0.05 are considered significant.

ELIGIBILITY:
Inclusion Criteria:

* emergency calls for epileptic seizures received by the emergency medical system of Zurich,Switzerland,
* the use of midazolam or diazepam or no drug used.

Exclusion Criteria:

* the use of any other first line drug to stop seizures than the two mentioned above e.g. thiopental

Max Age: 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: retrospective collected data from the emergency medical system "Schutz & Rettung Zürich", Zurich, Switzerland, over an 18 months period from 01. June 2013 till 31. December 2014 - all calls for epileptic seizures
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Which drug (Midazolam versus Diazepam) better stops epileptic seizures in the pre-clinical setting | follow up up to 1 year
  In this retrospective trial, all Emergency Medical Services of the city of Zurich interventions due to epileptic seizures during June 2013 and December 2014 are analyzed regarding the two drugs (Midazolam or Diazepam) used, its application mode (intravenous, nasal, intramuscular, rectal) and the application mode based success. Data will be collected regarding these aspects in order to determine if one drug is better than the other one, and which application mode is the most efficient.
  Furthermore, children versus adults are compared. Continuous variables are summarized as mean ± standard deviation (SD) and also presented as median [minimum; maximum]. Groups are compared using the independent samples t-test. P-values < 0.05 are considered significant.

SECONDARY OUTCOMES:
Does the way of application of the drugs (Midazolam versus Diazepam) used in pre-clinical epileptic seizures influence the outcome | follow up up to 1 year
  In this retrospective trial, all Emergency Medical Services of the city of Zurich interventions due to epileptic seizures during June 2013 and December 2014 are analyzed regarding the two drugs (Midazolam or Diazepam) used, its application mode (intravenous, nasal, intramuscular, rectal) and the application mode based success. Data will be collected regarding these aspects in order to determine if one drug is better than the other one, and which application mode is the most efficient.
  Furthermore, children versus adults are compared. Continuous variables are summarized as mean ± standard deviation (SD) and also presented as median [minimum; maximum]. Groups are compared using the independent samples t-test. P-values < 0.05 are considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver M Theusinger, MD, Study Chair — Balgrist University Hospital

IPD SHARING:
Plan to Share IPD: No